CLINICAL TRIAL: NCT00746876
Title: Unipolar or Bipolar Hemiarthroplasty in the Treatment of Displaced Femoral Neck Fractures. A Randomized Trial of RSA Measurements of Acetabular Wear.
Brief Title: Unipolar or Bipolar Hemiarthroplasty in the Treatment of Displaced Femoral Neck Fractures.
Acronym: HEMIUNIBIPOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Asker og Baerum (Other)
Collaborators: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Wender Figved, MD PhD, Sykehuset Asker og Baerum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMI-UNI-BIPOL
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Hip Fractures
Keywords: Hip; Fracture; Femoral neck; Hemiarthroplasty; Bipolar; Unipolar; Displaced femoral neck fractures
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unipolar (Active Comparator): 15 patients randomized for treatment with a unipolar hip hemiarthroplasty
  Interventions: Device: Unipolar hip hemiarthroplasty
- Bipolar (Active Comparator): 15 patients randomized for treatment with a bipolar hip hemiarthroplasty
  Interventions: Device: Bipolar hip hemiarthroplasty

INTERVENTIONS:
Device: Unipolar hip hemiarthroplasty — Unipolar hip hemiarthroplasty for the treatment of femoral neck fractures
  Other Names: Modular Cathcart Unipolar, DePuy/Johnson and Johnson
  Arms: Unipolar
Device: Bipolar hip hemiarthroplasty — Bipolar hip hemiarthroplasty for the treatment of femoral neck fractures
  Other Names: Celf-Centering Bipolar, DePuy/Johnson and Johnson
  Arms: Bipolar

SUMMARY:
Hemiarthroplasty of the hip is standard treatment of femoral neck fractures (hip fractures). Hemiarthroplasty means replacing the hip joint with a metal prosthesis. Unipolar prostheses has a one-piece design where the hip movement occurs between the prosthesis and the acetabulum (hip socket). A bipolar prosthesis has an additional artificial joint between the two components of the prosthesis. Both treatments are clinically proven and common around the world. No clinical trial has proven benefits of one or the other prosthesis design. The investigators want to measure the differences in acetabular wear using these two prostheses, using radiostereometric measurements.

DETAILED DESCRIPTION:
Patients 70 years or older presenting to our hospital with an acute femoral neck fracture are eligible for inclusion. 15 patients in each group will be recruited. One group receives a unipolar hemiarthroplasty and 15 receives a bipolar arthroplasty. Tantalum markers are placed around the acetabulum during surgery. Follow-up intervals are at 3, 12 and 24 months with radiostereometric evaluation (radiographs) and clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* 70 years or older
* Ambulatory status: No walking aids
* No mental illness or impaired cognitive function

Exclusion Criteria:

* Pathological fracture (malignant disease)
* Ongoing systemic or local infection
* Radiologically presence of acetabular wear (osteoarthrosis)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acetabular wear measured with radiostereometry | 24 months

SECONDARY OUTCOMES:
Harris hip score | 24 months
Health-related quality of life (eq-5d) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Hjall, M.D., Study Director — Asker and Baerum hospital, Norway
Locations (1):
- Asker and Baerum Hospital, Baerum, Rud, Norway